CLINICAL TRIAL: NCT03783897
Title: A Phase 1, Open-label, Fixed-sequence Study to Investigate the Effects of EDP 305 on the Pharmacokinetics of a Combined Oral Contraceptive in Healthy Adult Female Subjects
Brief Title: A Drug-drug Interaction Study to Investigate the Effect of Coadministration of EDP-305 on the PK of a Combined Oral Contraceptive in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 305-008
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
Keywords: OC DDI, drug-drug interaction, oral contraceptive
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — EDP-305; Contraceptives, Oral; Ethinyl Estradiol; norgestimate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EDP-305 and Oral Contraceptive (Experimental)
  Interventions: Drug: EDP-305; Drug: Oral Contraceptive

INTERVENTIONS:
Drug: EDP-305 — Subjects will receive EDP-305 on on Days 11 through 21 of cycle 3
Drug: Oral Contraceptive — Subjects will receive active Oral Contraceptive on Days 1-21 and inert OC on Days 22-28 of cycles 1, 2 and 3
  Other Names: ethinyl estradiol [EE] and norgestimate [NGM])

SUMMARY:
A Phase 1, Open-label, Fixed-sequence Study to Investigate the Effects of EDP 305 on the Pharmacokinetics of a Combined Oral Contraceptive in Healthy Adult Female Subjects

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential, 18 to 45 years of age, inclusive. Follicle-stimulating hormone levels may be used to confirm premenopausal status, including females who have had a hysterectomy with ovaries still intact. Women who otherwise meet inclusion criteria and who have had tubal ligation, tubal occlusion, or bilateral salpingectomy will be allowed.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations at Screening and Day -1 of the Lead-in Period
* Must not be pregnant or lactating, and must agree to use contraception
* Subjects must have documentation of normal results of up-to-date cervical cancer screening as specified in the American College of Obstetricians and Gynecologists guidelines:

  1. Women aged < 21 years: no documentation required
  2. Women aged 21 to 29: normal Pap smear test result within previous 3 years
  3. Women aged 30 to 45: normal Pap smear test result and negative high-risk human papilloma virus test within previous 5 years, OR normal Pap smear test result within previous 3 years If documented results are not available at Screening, the subject must provide documentation of normal results prior to Day -1 of the Lead-in Period.
* Able to comprehend and willing to sign an ICF.
* Willing and able to adhere to assessments, prohibitions, and restrictions as described in this protocol.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, GI, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* Are pregnant, breastfeeding, or are planning to conceive during the study.
* Have been administered injectable contraceptives within 12 months prior to Day -1 of the Lead in Period, or had exposure to a hormonal intrauterine device or topical controlled delivery contraceptives (patch) within 3 months prior to Day -1 of the Lead-in Period.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 43 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time (AUC0-τ) curve for OC with and without coadministration with EDP-305 | Day 21 (cycle 2 and cycle 3)
Cmax for OC with and without coadministration with EDP-305 | Day 21 (cycle 2 and cycle 3)

SECONDARY OUTCOMES:
Area under the plasma concentration-time (AUC0-τ) curve for EDP-305 when coadministration with OC | Days 14, 20-22 (cycle 3)
Cmax for EDP-305 when coadministration with OC | Days 14, 20-22 (cycle 3)
Safety measured by adverse events | Approximately 91 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States